CLINICAL TRIAL: NCT06319716
Title: LINK-IT: Leveraging Videos and Community Health Workers to Address Social Determinants of Health in Immigrants
Brief Title: Leveraging Videos and Community Health Workers to Address Social Determinants of Health in Immigrants
Acronym: LINK-IT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 23-01274
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Palliative Care; Community Health Workers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VIDEO (Experimental): Participants assigned to the VIDEO arm will receive one brief Diabetes Self-Management Education and Support (DSMES) video per week for 24 weeks. The videos will be delivered via text message.
  Interventions: Behavioral: Video-Based Diabetes Self-Management Education and Support (DSMES)
- VIDEO+CHW (Experimental): Participants assigned to the VIDEO+CHW arm will receive one brief DSMES video per week, in addition to bi-weekly support calls from a community health worker (CHW), for 24 weeks. The DSMES videos will be delivered via text message.
  Interventions: Behavioral: Video-Based Diabetes Self-Management Education and Support (DSMES); Behavioral: Community Health Worker (CHW) Support
- CONTROL (No Intervention): Participants assigned to the CONTROL group will continue to receive usual care.

INTERVENTIONS:
Behavioral: Video-Based Diabetes Self-Management Education and Support (DSMES) — The DSMES videos provide important diabetes education to participants and empower them to become an activated patient on the individual level.
  Arms: VIDEO; VIDEO+CHW
Behavioral: Community Health Worker (CHW) Support — CHWs will assess participants' social determinants of health (SDOH) barriers to Type 2 diabetes care and link them to available resources in the community.
  Arms: VIDEO+CHW

SUMMARY:
The overall goal of this study is to examine the efficacy of the video-based Diabetes Self-Management Education and Support (DSMES) (hereafter VIDEO), or the video-based DSMES+community health worker (CHW) intervention (hereafter VIDEO+CHW), compared with a wait-list control group (hereafter CONTROL) to improve glycemic control among Chinese immigrants with uncontrolled Type 2 diabetes in NYC.

DETAILED DESCRIPTION:
Participants will be randomized with equal allocation to one of the 3 groups. The VIDEO group will receive 1 DSMES brief video/week for 24 weeks delivered via text message. The VIDEO+CHW group will receive the same DSMES videos plus bi-weekly support calls from a CHW for 24 weeks. The CHW will assess participants' social determinants of health (SDOH) barriers to Type 2 diabetes care and link them to available resources in the community. The CONTROL group will continue to receive their usual care and at the end of the study, they will receive DSMES videos.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as a Chinese immigrant;
* be above 18 years old;
* have a diagnosis of Type 2 diabetes (T2D) in the medical record;
* have had an appointment with a physician for routine T2D care within the past 12 months;
* have a most recent HbA1c of at least 7%;
* be willing to receive brief videos regarding T2D management; and
* possess a smartphone or, if they do not have one, be willing and able to use a study smartphone.

Exclusion Criteria:

* unable or unwilling to provide informed consent;
* unable to participate meaningfully in the intervention (e.g., uncorrected sight and hearing impairment);
* unwilling to accept randomization assignment;
* is pregnant, plans to become pregnant in the next 6 months, or becomes pregnant during the study; or
* is breastfeeding (e.g., they may have potential dietary restrictions).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-12-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c (HbA1c) Levels | Baseline
Hemoglobin A1c (HbA1c) Levels | Month 6
Hemoglobin A1c (HbA1c) Levels | Month 12

SECONDARY OUTCOMES:
Stanford Self-Efficacy for Diabetes Scale Score | Baseline
  8-item self-assessment of participants' confidence level in performing specific self-management behaviors. Items are ranked on a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident). The total score is the average of all scores and ranges from 1-10; where higher scores indicate greater self-efficacy.
Stanford Self-Efficacy for Diabetes Scale Score | Month 6
  8-item self-assessment of participants' confidence level in performing specific self-management behaviors. Items are ranked on a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident). The total score is the average of all scores and ranges from 1-10; where higher scores indicate greater self-efficacy.
Stanford Self-Efficacy for Diabetes Scale Score | Month 12
  8-item self-assessment of participants' confidence level in performing specific self-management behaviors. Items are ranked on a 10-point Likert scale ranging from 1 (not at all confident) to 10 (totally confident). The total score is the average of all scores and ranges from 1-10; where higher scores indicate greater self-efficacy.
Starting the Conversation (STC) Diet Scale Score | Baseline
  8-item self-report questionnaire measuring dietary behaviors. Scores range from 0 to 16; lower scores indicate more dietary behaviors that are consistent with health.
Starting the Conversation (STC) Diet Scale Score | Month 6
  8-item self-report questionnaire measuring dietary behaviors. Scores range from 0 to 16; lower scores indicate more dietary behaviors that are consistent with health.
Starting the Conversation (STC) Diet Scale Score | Month 12
  8-item self-report questionnaire measuring dietary behaviors. Scores range from 0 to 16; lower scores indicate more dietary behaviors that are consistent with health.
International Physical Activity Questionnaire (IPAQ) Short-Version Score | Baseline
  Self-assessment providing an estimate of the number of minutes per week participants engage in three categories of physical activity: vigorous activity, moderate activity, and walking activity. Results are expressed in metabolic equivalent (MET) minutes per week. MET minutes represent the amount of energy expended carrying out physical activity. The formula for calculating MET is as follows: 8(vigorous activity)(minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes) = MET.
  Higher MET scores indicate higher weekly levels of physical activity.
International Physical Activity Questionnaire (IPAQ) Short-Version Score | Month 6
  Self-assessment providing an estimate of the number of minutes per week participants engage in three categories of physical activity: vigorous activity, moderate activity, and walking activity. Results are expressed in metabolic equivalent (MET) minutes per week. MET minutes represent the amount of energy expended carrying out physical activity. The formula for calculating MET is as follows: 8(vigorous activity)(minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes) = MET.
  Higher MET scores indicate higher weekly levels of physical activity.
International Physical Activity Questionnaire (IPAQ) Short-Version Score | Month 12
  Self-assessment providing an estimate of the number of minutes per week participants engage in three categories of physical activity: vigorous activity, moderate activity, and walking activity. Results are expressed in metabolic equivalent (MET) minutes per week. MET minutes represent the amount of energy expended carrying out physical activity. The formula for calculating MET is as follows: 8(vigorous activity)(minutes) + 4 (moderate activity)(minutes) +3.3 (walking activity) (minutes) = MET.
  Higher MET scores indicate higher weekly levels of physical activity.
Adherence to Refills and Medications Scale for Diabetes (ARMS-D) | Baseline
  ARMS-D is an 11-item questionnaire used to assess medication-taking adherence at baseline, 6 months, and 12 months. Responses range from 1 ("none of the time") to 4 ("all of the time"). Item scores are summed to produce an overall adherence score ranging from 12 to 48, with higher scores indicating more problems with medication adherence.
Adherence to Refills and Medications Scale for Diabetes (ARMS-D) | Month 6
  ARMS-D is an 11-item questionnaire used to assess medication-taking adherence at baseline, 6 months, and 12 months. Responses range from 1 ("none of the time") to 4 ("all of the time"). Item scores are summed to produce an overall adherence score ranging from 12 to 48, with higher scores indicating more problems with medication adherence.
Adherence to Refills and Medications Scale for Diabetes (ARMS-D) | Month 12
  ARMS-D is an 11-item questionnaire used to assess medication-taking adherence at baseline, 6 months, and 12 months. Responses range from 1 ("none of the time") to 4 ("all of the time"). Item scores are summed to produce an overall adherence score ranging from 12 to 48, with higher scores indicating more problems with medication adherence.
Emotional Support Subscale from the NIH Toolbox Adult Social Relationship Scales | Baseline
  8-item subscale to assess individuals' perceptions of empathy and understanding received from others in their social network at baseline, 6 months, and 12 months. Total scores range from 8 to 40, with higher scores indicating greater perceived emotional support.
Emotional Support Subscale from the NIH Toolbox Adult Social Relationship Scales | Month 6
  8-item subscale to assess individuals' perceptions of empathy and understanding received from others in their social network at baseline, 6 months, and 12 months. Total scores range from 8 to 40, with higher scores indicating greater perceived emotional support.
Emotional Support Subscale from the NIH Toolbox Adult Social Relationship Scales | Month 12
  8-item subscale to assess individuals' perceptions of empathy and understanding received from others in their social network at baseline, 6 months, and 12 months. Total scores range from 8 to 40, with higher scores indicating greater perceived emotional support.

CONTACTS AND LOCATIONS:
Overall Officials: Lu Hu, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Lu.hu@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Lu.hu@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Hu L, Liu J, Yang X, Teng C, Li H, Zhao Y, Levy N, Zhu K, Vang S, Kwon SC, Feldman N, Lau J, Jiang Y, Trinh-Shevrin C, Islam N. Leveraging videos and community health workers to address social determinants of health in immigrants (LINK-IT): Protocol for a randomized controlled trial. PLoS One. 2026 Feb 2;21(2):e0341217. doi: 10.1371/journal.pone.0341217. eCollection 2026. PMID 41628090